CLINICAL TRIAL: NCT04595578
Title: Effect of Repetitive Transcranial Magnetic Stimulation With Intensive Physical Therapy in Cerebellar Ataxia: A Pilot Study
Brief Title: Cerebellar rTMS and Physical Therapy for Cerebellar Ataxia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Jinyoung Youn, Associate Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2017-10-166
Record Dates: First submitted 2020-10-07; First posted 2020-10-20 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-10

CONDITIONS: Multiple System Atrophy, Cerebellar Variant (Disorder); Spinocerebellar Ataxias
MeSH Terms: conditions — Multiple System Atrophy; Spinocerebellar Ataxias

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cerebellar rTMS + Physical therapy (Active Comparator): rTMS was delivered on the scalp for over 2 cm under the inion, which is the scalp over the cerebellum area, using a double-cone coil connected to a Magstim Rapid2® stimulator with two Booster Modules (Magstim, Spring Gardens, Wales, UK) in accordance with safety recommendations. Stimulation was delivered to the cerebellum at 10 Hz with 90% of the mean resting motor threshold intensity for 5 seconds at 55 second intervals to deliver 1000 pulses in 20 minutes. Immediately after rTMS, the combination treatment group received balance and gait training by a physical therapist for 30 minutes/day and underwent aerobic exercise using a stationary bicycle at moderate intensity (12 to 14 rating of perceived exertion) for 30 minutes/day and 5 days/week for two weeks. In the control group, no participants received physical therapy or rTMS for two weeks.
  Interventions: Device: Cerebellar repetitive transcranial magnetic stimulation
- Sham stimulation + Physical therapy (Sham Comparator): Sham stimulation was delivered on the scalp for over 2 cm under the inion, which is the scalp over the cerebellum area, using a double-cone coil connected to a Magstim Rapid2® stimulator. Sham stimulation was delivered to the cerebellum for 5 seconds at 55 second intervals in 20 minutes. Immediately after rTMS, the combination treatment group received balance and gait training by a physical therapist for 30 minutes/day and underwent aerobic exercise using a stationary bicycle at moderate intensity (12 to 14 rating of perceived exertion) for 30 minutes/day and 5 days/week for two weeks. In the control group, no participants received physical therapy or rTMS for two weeks.
  Interventions: Device: Cerebellar repetitive transcranial magnetic stimulation

INTERVENTIONS:
Device: Cerebellar repetitive transcranial magnetic stimulation — rTMS was delivered on the scalp for over 2 cm under the inion, which is the scalp over the cerebellum area, using a double-cone coil connected to a Magstim Rapid2® stimulator with two Booster Modules (Magstim, Spring Gardens, Wales, UK) in accordance with safety recommendations. Stimulation was delivered to the cerebellum at 10 Hz with 90% of the mean resting motor threshold intensity for 5 seconds at 55 second intervals to deliver 1000 pulses in 20 minutes. Immediately after rTMS, the combination treatment group received balance and gait training by a physical therapist for 30 minutes/day and underwent aerobic exercise using a stationary bicycle at moderate intensity (12 to 14 rating of perceived exertion) for 30 minutes/day and 5 days/week for two weeks. In the control group, no participants received physical therapy or rTMS for two weeks.

SUMMARY:
The present study investigated the efficacy and safety of combination treatment of repetitive transcranial magnetic stimulation (rTMS) and physical therapy (PT) in patients with cerebellar variant of multiple system atrophy (MSA-C) and spinocerebellar ataxia.

ELIGIBILITY:
Inclusion Criteria:

1. The patients with probable MSA-C and spinocerebellar ataxia (SCA)
2. cerebellar ataxia as main clinical presenting feature and able to walk independently without walking devices
3. aged over 20
4. presence of cerebellar atrophy proven by brain MRI.

Exclusion Criteria:

1. secondary cerebellar ataxia
2. peripheral neuropathy, radiculopathy, or decreased visual acuity that can cause peripheral ataxia
3. musculoskeletal disease affecting gait or balance
4. other neurologic symptoms, including symptomatic parkinsonism (two or more rigidity and/or bradykinesia scores in one limb by Unified Parkinson's disease Rating Scale part 3) or spasticity (20)
5. psychiatric symptoms requiring medication or with cognitive decline (Mini-mental state examination [MMSE] < 20)
6. taking any sedative medications or anti-parkinsonian medications such as benzodiazepine, levodopa or dopamine agonist
7. history of seizure or metallic brain implants; (8) cardiopulmonary diseases causing dyspnea during exercise.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
International Cooperative Ataxia Rating Scale (ICARS) | The change of ICARS score between baseline (T0) and immediately after (T1) treatment
  The scale is scored out of 100 with 19 items and 4 subscales of postural and gait disturbances, limb ataxia, dysarthria, and oculomotor disorders. Higher scores indicate higher levels of impairment.

SECONDARY OUTCOMES:
Change from temporospatial parameters of gait | The clinical scales were evaluated by blinded raters at baseline (T0) and immediately after (T1), 4 weeks after (T2), and 12 weeks (T3) after intervention.
  Gait parameters measured by GAITRite system
Change from posturography | The clinical scales were evaluated by blinded raters at baseline (T0) and immediately after (T1), 4 weeks after (T2), and 12 weeks (T3) after intervention.
  Posturography measured by Pedoscan system
Change from Mini-Mental State Examination (MMSE) | The clinical scales were evaluated by blinded raters at baseline (T0) and immediately after (T1), 4 weeks after (T2), and 12 weeks (T3) after intervention.
  Measurement of cognitive function
Change from Beck depression inventory (BDI) | The clinical scales were evaluated by blinded raters at baseline (T0) and immediately after (T1), 4 weeks after (T2), and 12 weeks (T3) after intervention.
  Measurement of symptoms of depression
Change from Barthel Index for Activities of Daily Living | The clinical scales were evaluated by blinded raters at baseline (T0) and immediately after (T1), 4 weeks after (T2), and 12 weeks (T3) after intervention.
  Measurement of activities of daily living
Change from International Cooperative Ataxia Rating Scale (ICARS) | The clinical scales were evaluated by blinded raters at baseline (T0) and 4 weeks after (T2), and 12 weeks (T3) after intervention.
  The scale is scored out of 100 with 19 items and 4 subscales of postural and gait disturbances, limb ataxia, dysarthria, and oculomotor disorders. Higher scores indicate higher levels of impairment.

CONTACTS AND LOCATIONS:
Overall Officials: Jong Hyeon Ahn, Study Director — Samsung Medical Center, Department of Neurology
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No